CLINICAL TRIAL: NCT00217451
Title: Evaluation of Fosmidomycin in Combination With Clindamycin in Children With Acute Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Treatment of Malaria in Gabon With Fosmidomycin-Clindamycin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Schweitzer Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06/2002/FOS-CLIN/JP006
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Malaria
Keywords: Malaria; Fosmidomycin; Clindamycin; Gabon
MeSH Terms: conditions — Malaria

INTERVENTIONS:
Drug: Fosmidomycin-clindamycin

SUMMARY:
Some antibiotics are also effective against malaria parasites. Fosmidomycin is an antibiotic that has been shown to be effective against malaria, although it cannot achieve a total cure in all patients. A previous small study has shown that in combination with clindamycin, an commonly used antibiotic, it is highly effective and safe, in asymptomatic carriers of malaria parasites. The current study will evaluate the efficacy and safety of the combination given for three days in children with uncomplicated malaria in Gabon.

DETAILED DESCRIPTION:
The treatment of malaria is becoming increasingly difficult due to the development of Plasmodium falciparum strains resistant to commonly used antimalarials. Fosmidomycin was shown to be well tolerated and fast-acting in paediatric outpatients and adults, but late recrudescences preclude its use as monotherapy. Clindamycin was identified as a suitable combination partner following the demonstration of synergistic inhibition of plasmodial growth by in vitro and animal studies.

In this study, the safety and efficacy of fosmidomycin-clindamycin (30 mg/kg plus 10 mg/kg) twice daily for three days is assessed in children with acute uncomplicated P. falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated P. falciparum malaria with acute manifestation
* Asexual parasitemia between 1,000-100,000/μL
* Body weight between 5-65 kg
* Ability to tolerate oral therapy
* Informed consent, oral agreement of the child if appropriate
* Residence in the study area for the duration of at least 4 weeks

Exclusion Criteria:

* Adequate anti-malarial treatment within the previous 7 days
* Antibiotic treatment for a concurrent infection
* Haemoglobin <7g/dL
* Hematocrit <25%
* Leukocyte count >15,000/μL
* Mixed plasmodial infection
* Severe malaria, any other severe underlying disease
* Concomitant disease masking assessment of treatment response
* Inflammatory bowel disease, and any other disease causing fever.

Ages: 12 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51
Dates: Start 2002-06; Study Completion 2003-03

PRIMARY OUTCOMES:
Proportion of patients cured by day 14
Incidence of adverse events after the start of treatment

SECONDARY OUTCOMES:
Parasite clearance time
Fever clearance time
PCR corrected day 28 cure rate

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Borrmann, MD, Principal Investigator — Kenya Medical Research Institute, Centre for Geographic Medicine Research, Coast, kilifi, Kenya; Peter G. Kremsner, MD, FRCP, Principal Investigator — Albert Schweitzer Hospital
Locations (1):
- Medical Research Unit, Lambaréné, Lambaréné, Moyen-Ogooué Province, Gabon

REFERENCES:
- [Background] Beytia ED, Porter JW. Biochemistry of polyisoprenoid biosynthesis. Annu Rev Biochem. 1976;45:113-42. doi: 10.1146/annurev.bi.45.070176.000553. No abstract available. PMID 9026
- [Background] Lois LM, Campos N, Putra SR, Danielsen K, Rohmer M, Boronat A. Cloning and characterization of a gene from Escherichia coli encoding a transketolase-like enzyme that catalyzes the synthesis of D-1-deoxyxylulose 5-phosphate, a common precursor for isoprenoid, thiamin, and pyridoxol biosynthesis. Proc Natl Acad Sci U S A. 1998 Mar 3;95(5):2105-10. doi: 10.1073/pnas.95.5.2105. PMID 9482846
- [Background] Rohmer M, Knani M, Simonin P, Sutter B, Sahm H. Isoprenoid biosynthesis in bacteria: a novel pathway for the early steps leading to isopentenyl diphosphate. Biochem J. 1993 Oct 15;295 ( Pt 2)(Pt 2):517-24. doi: 10.1042/bj2950517. PMID 8240251
- [Background] Jomaa H, Wiesner J, Sanderbrand S, Altincicek B, Weidemeyer C, Hintz M, Turbachova I, Eberl M, Zeidler J, Lichtenthaler HK, Soldati D, Beck E. Inhibitors of the nonmevalonate pathway of isoprenoid biosynthesis as antimalarial drugs. Science. 1999 Sep 3;285(5433):1573-6. doi: 10.1126/science.285.5433.1573. PMID 10477522
- [Background] Clinical study report for Protocol JP 001 - Evaluation of fosmidoymcin in adult patients with acute uncomplicated Plasmodium falciparum malaria. 2001. World Health Organisation, Geneva, Switzerland and Jomaa Pharmaka GmbH, Germany
- [Background] Wiesner J, Henschker D, Hutchinson DB, Beck E, Jomaa H. In vitro and in vivo synergy of fosmidomycin, a novel antimalarial drug, with clindamycin. Antimicrob Agents Chemother. 2002 Sep;46(9):2889-94. doi: 10.1128/AAC.46.9.2889-2894.2002. PMID 12183243
- See also: General information on malaria at the website of the Malaria Foundation International — http://www.malaria.org
- See also: Homepage of Medical Research Unit, Lambaréné — http://www.lambarene.org